CLINICAL TRIAL: NCT00881231
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Eon and Otsuka (Pletal) 50 mg Cilostazol Tablets In Healthy Adults Volunteers Under Fasting Conditions
Brief Title: To Demonstrate the Relative Bioavailability of Cilostazol 50 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA17524
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Cilostazol; Long-Term Synaptic Depression

ARMS (2):
- 1 (Experimental): Cilostazol 50 mg Tablets (Eon Pharma, LLC, USA)
  Interventions: Drug: Cilostazol 50 mg Tablets (Eon Pharma, LLC, USA)
- 2 (Active Comparator): Pletal (Cilostazol) 50 mg Tablets (Otsuka Pharma Co, Ltd., USA)
  Interventions: Drug: Pletal (Cilostazol) 50 mg Tablets (Otsuka Pharma Co, Ltd., USA)

INTERVENTIONS:
Drug: Cilostazol 50 mg Tablets (Eon Pharma, LLC, USA)
  Arms: 1
Drug: Pletal (Cilostazol) 50 mg Tablets (Otsuka Pharma Co, Ltd., USA)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability of Cilostazol 50 mg tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2004-01; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, M.D., Principal Investigator — MDS Pharma Services